# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Initial Evaluation of Investigational Lenses Manufactured on a New Production Line

Protocol: CR-6283

Version: 3.0, Amendment 2.0

Date: 09 Aug 2018

Investigational Products: Senofilcon-based contact lens containing new-UV blocker

Key Words: senofilcon A, Subjective Performance, Fitting Characteristics, Dispensing, Daily

Wear

# Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>1</sup> ISO 14155,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

## **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# TABLE OF CONTENTS PROTOCOL TITLE, NUMBER, VERSION.....6 SPONSOR NAME AND ADDRESS......6 MEDICAL MONITOR......6 AUTHORIZED SIGNATURES.......7 CHANGE HISTORY......8 SYNOPSIS.......9 COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS ......14 1.1. 1.2. 1.3. 1.4. 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES .......17 2.1. 2.2. 2.3. 3. TARGETED STUDY POPULATION .......22 3.1. 3.2. Inclusion Criteria 23 3.3. Exclusion Criteria 23 3.4. 4. STUDY DESIGN AND RATIONALE.....24 Description of Study Design ......24 4.1. 4.2. Study Design Rationale .......25 4.3. 5. TEST ARTICLE ALLOCATION AND MASKING.......25 5.1. 5.2. 5.3. Procedures for Maintaining and Breaking the Masking......26 6.1. 6.2. Ancillary Supplies/Products......27

| 6.3. | Administration of Test Articles | 27 |
|---|---|---|
| 6.4. | Packaging and Labeling | 28 |
| 6.5. | Storage Conditions | 28 |
| 6.6. | Collection and Storage of Samples | 28 |
| 6.7. | Accountability of Test Articles | 28 |
| 7. ST | UDY EVALUATIONS | 30 |
| 7.1. | Time and Event Schedule | 30 |
| 7.2. | Detailed Study Procedures | 31 |
| VI | ISIT 1 | 31 |
| VI | ISIT 2 | 35 |
| VI | ISIT 3 | 39 |
| VI | ISIT 4 | 44 |
| FI | NAL EVALUATION | 46 |
| 7.3. | Unscheduled Visits | 46 |
| 7.4. | Laboratory Procedures | 48 |
| 8. SU | BJECTS COMPLETION/WITHDRAWAL | |
| 8.1. | Completion Criteria | 48 |
| 8.2. | Withdrawal/Discontinuation from the Study | 48 |
| 9. PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 49 |
| 10. DE | VIATIONS FROM THE PROTOCOL | 49 |
| 11. ST | UDY TERMINATION | 49 |
| 12. PR | OCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 50 |
| 13. AD | OVERSE EVENTS | 51 |
| 13.1. | Definitions and Classifications | 51 |
| 13.2. | Assessing Adverse Events | 53 |
| 13 | 3.2.1 Causality Assessment | 53 |
| 13 | 3.2.2 Severity Assessment | 54 |
| 13.3. | Documentation and Follow-Up of Adverse Events | 54 |
| 13.4. | Reporting Adverse Events | 55 |
| 13 | 3.4.1 Reporting Adverse Events to Sponsor | 55 |
| 13 | 3.4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Aut | thorities.56 |
| 13.4. | 3 Event of Special Interest | 56 |
| 13.5. | Reporting of Pregnancy | 57 |
| 14. ST | ATISTICAL METHODS | 57 |

| 14.1. General Considerations | 57 |
|---|---|
| 14.2. Sample Size Justification. | 57 |
| 14.3. Analysis Populations | 62 |
| 14.4. Level of Statistical Significance | 63 |
| 14.5. Primary Analysis | 63 |
| 14.6. Secondary Analysis | 69 |
| 14.7. Other Exploratory Analyses | 69 |
| 14.8. Interim Analysis | 70 |
| 14.9. Procedure for Handling Missing Data and Drop-Outs | 70 |
| 14.10. Procedure for Reporting Deviations from Statistical Plan | 70 |
| 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING | 70 |
| 15.1. Electronic Case Report Form/Data Collection | 70 |
| 15.2. Subject Record | 71 |
| 16. DATA MANAGEMENT | 71 |
| 16.1. Access to Source Data/Document | 71 |
| 16.2. Confidentiality of Information | 72 |
| 16.3. Data Quality Assurance | 72 |
| 17. MONITORING | 72 |
| 18. ETHICAL AND REGULATORY ASPECTS | 73 |
| 18.1. Study-Specific Design Considerations | 73 |
| 18.2. Investigator Responsibility | 73 |
| 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 73 |
| 18.4. Informed Consent | 74 |
| 18.5. Privacy of Personal Data | 75 |
| 19. STUDY RECORD RETENTION | 76 |
| 20. FINANCIAL CONSIDERATIONS | 76 |
| 21. PUBLICATION | 77 |
| 22. REFERENCES | 78 |
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 79 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | 104 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APPENDIX D: CLINICAL TECHNICAL PROCEDURES | 108 |
| LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS | 109 |
| EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 117 |

| LENS FITTING CHARACTERISTICS | 122 |
|---|---|
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | 129 |
| FRONT AND BACK SURFACE LENS DEPOSIT GRADING | |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL RI | |
| BIOMICROSCOPY SCALE | 144 |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 150 |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT | |
| PATIENT REPORTED OUTCOMES | |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILL<br>TESTING | |
| qCSF CONTRAST SENSITIVITY | 167 |
| APPENDIX E: IRIS COLOR | 174 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 176 |
| TABLE OF CONTENTS | |
| Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | 27 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |
| Table 5: Descriptive Summary of CLUE Scores by Domain Pooled Across His | |
| ) – 2-Week Follow-up Evaluation | 58 |
| Table 6: Descriptive Summary of Visual Acuity (logMAR) 2-W | |
| Evaluation | storical Studies |
| Table 8: Descriptive Summary of Slit Lamp Findings Pooled Across all Histor. Table 9: Descriptive Summary of Individual Items from ———————————————————————————————————— | ical Studies 59<br>ollow-up 60<br>ts62 |
| Table 11: Sample Size Estimates and Power Calculations for Secondary Endpo | oints |

# PROTOCOL TITLE, NUMBER, VERSION

Title: Initial Evaluation of Investigational Lenses Manufactured on a New Production Line

Protocol Number: CR-6283 Version: 3.0, Amendment 2.0

Date: 09 August 2018

## SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway, Jacksonville, FL 32256

## **MEDICAL MONITOR**

Name: John R. Buch, O.D., M.S., F.A.A.O. Title: Principal Research Optometrist Address:

Email: jbuch@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

## **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>1</sup> ISO 14155<sup>2</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Report Name: John R. Buch, O.D., M.S. Title: Principal Research Optometrist | DATE |
|---|---|---|
| Clinical Operations | | |
| Manager | See Electronic Signature Report Name: Title: Clinical Operations Manager | DATE |
| Biostatistician | See Electronic Signature Report | |
| | Name: Title: Biostatistician II | DATE |
| Biostatistician | | |
| Reviewer | See Electronic Signature Report Name: Title: Manager of Biostatistics | DATE |
| Reviewer | See Electronic Signature Report | |
| | Name: Title: Clinical Research Fellow | DATE |
| Data Management | See Electronic Signature Report Name: Title: Clinical Project Manager, Data and Systems | DATE |
| Approver | See Electronic Signature Report Name: Title: Reusable Platform Lead | DATE |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | John Buch | Original Protocol | 01 August 2018 |
| 2.0 | John Buch | Updated 'Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them,' to an individual inclusion criteria. Moved Inclusion Criteria after Baseline # 7-10 to Inclusion Criteria after Screening. Moved Exclusion Criteria after Baseline # 13-14 to Exclusion Criteria After Screening | 07 August 2018 |
| 3.0 | John Buch | Update 'The subject must have visual acuity best correctable to 20/25+3 or better for each eye.' To an individual inclusion criteria | 09 August 2018 |

# **SYNOPSIS**

| Protocol Title | Initial Evaluation of Investigational Lenses Manufactured on a New Production Line |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development Phase 2b |
| Trial Registration | This study will be registered on ClinicalTrials.gov |
| Test Article(s) | Investigational Products: Senofilcon-based contact lens containing new-UV blocker (Test lens) |
| | Control Products: Commercial ACUVUE® OASYS® |
| Wear and Replacement | Wear Schedule: daily wear (DW) |
| Schedules | Replacement Schedule: approximately 2 weeks |
| Objectives | The primary objective of this study is to demonstrate non-inferiority of the Test lens compared to the Control lens with respect to CLUE comfort, Slit Lamp Findings and Monocular Distance Visual Acuity (logMAR). This study will also aim to show the Fit Acceptance rate of the Test lens is at least 90%. |
| Study Endpoints | Primary Endpoints: |
| | <ul> <li>Monocular distance visual acuity (logMAR)</li> <li>Slit Lamp Findings (Grade 3 or Higher)</li> <li>Fit acceptance rate</li> <li>Overall CLUE comfort</li> </ul> |
| | Vision satisfaction in bright lighting |
| | Secondary Endpoints: |
| | <ul><li>Overall CLUE vision</li><li>Overall CLUE handling</li></ul> |
| Study Design | This study is a randomized, 4-visit, partially subject-masked, 2×3 bilateral crossover, dispensing trial. The study lenses will be worn as DW for a period of 2 weeks each with one of the study lenses being worn twice. Each study lens is expected to be worn at least five (5) days per week for at least six (6) hours per day. There will be no washout period between study lenses. There will be an interim analysis after 100 or more subjects have completed the first wearing period (2-weeks after initial lens dispensing). See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). |

| Sample Size | Approximately 120 eligible subjects will be enrolled and randomized into the study with a target of approximately 105 subjects to complete the study. A replacement subject may be enrolled if a subject discontinues from the study prematurely; the decision whether to enroll replacement subjects will be made by the joint agreement of the Investigator and Sponsor. |
|---|---|
| Study Duration | Subjects will wear the Test and Control lenses for 2 weeks each in random order with one of the study lenses being worn twice for a total of 6 weeks per subject. The enrollment period will be 2 weeks, making the entire study approximately 8 weeks in duration. |
| Anticipated Study Population | Approximately 120 subjects will be enrolled to ensure that at least 105 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of ≥18 and ≤49 years. |
| Eligibility Criteria (Inclusion Criteria) | <ol> <li>Potential subjects must satisfy all of the following inclusion criteria to be enrolled in the study: <ol> <li>The subject must read and sign the Informed Consent form.</li> <li>The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Healthy adult males or females age ≥18 and ≤49 years of age with signed informed consent.</li> <li>Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them</li> <li>The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and -6.00 D.</li> <li>The subject's refractive cylinder must be ≤ 1.00 D in each eye.</li> <li>Subjects must have visual acuity best correctable to 20/25<sup>+3</sup> or better for each eye.</li> <li>Subjects must own a wearable pair of spectacles.</li> <li>The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.</li> <li>Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week</li> <li>The subject must have normal eyes (i.e., no ocular medications or infections of any type).</li> </ol> </li> </ol> |

# Eligibility Criteria (Exclusion Criteria)

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
- 2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g., Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
- 4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
- 5. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 6. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g.., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
- 7. Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.
- 8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
- 9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.

| | <ul> <li>10. Toric, extended wear, monovision or multi-focal contact lens correction.</li> <li>11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.</li> <li>12. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.</li> <li>13. History of binocular vision abnormality or strabismus.</li> <li>14. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).</li> </ul> |
|---|---|
| Disallowed Medications/Interventions | Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication |
| Measurements and Procedures | Monocular distance visual acuity on logMAR scale using ETDRS charts, physiological responses, lens fitting characteristics, individual performance metrics, CLUE comfort, vision and handling. |
| Microbiology or Other<br>Laboratory Testing | The optical bench will be used to measure the light transmission characteristics for all worn test lenses. The findings are for internal information only and will not be part of the final report. |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the Control lens of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Opti-Free® PureMoist®, Preservative free rewetting drops/artificial tears |
| Principal Investigator(s)<br>and Study<br>Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



## COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee

DW Daily Wear

eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Council for Harmonization
IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

logMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator

PIG Patient Instruction Guide PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation SLF Slit Lamp Findings

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity UV Ultraviolet

HEV High energy visible

#### 1. INTRODUCTION AND BACKGROUND

ACUVUE® OASYS Transitions with Light Intelligent Technology was approved by the FDA in April 2018. The contact lenses will be produced on a new manufacturing line and clinically evaluated for the first time in this study.

## 1.1. Name and Descriptions of Investigational Products

Senofilcon-based contact lens containing a new-UV blocker.

## 1.2. Intended Use of Investigational Products

The intended use of the investigative product in this study is for correcting myopia and providing visual benefits in lighting situations where UV-A and/or High Energy Visible (HEV) light is present in the environment. During the study, each test article will be worn bilaterally in a daily wear (DW) modality for at least 6 hours per day and 5 days per week for approximately 2 weeks each. The subject will wear either the Test or Control article twice and the other study article once.

# 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding senofilcon A - based soft contact lens containing the new UV-blocker, refer to the latest version of the Investigator's Brochure for this study.

# 1.4. Known Risks and Benefits to Human Subjects

The risks of wearing soft contact lenses are well known and are described in the Investigator's Brochure and Informed Consent. The material safety testing/lens release criteria was determined based on the Risk Assessment.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Prior clinical data is summarized in the Investigator's Brochure.

The literature is absent of any articles pertaining to soft contact lenses containing the new type of UV-blocker. A list of relevant literature references pertaining to glare, eyestrain, and light filtering is provided:

- 1. Agarwal S, Goel D, Sharma A. Evaluation of the factors which contribute to the ocular complaints in computer users. *J Clin Diagn Res*. 2013;7(2):331-335.
- 2. Eperjesi F, Fowler CW, Evans BJ. Do tinted lenses or filters improve visual performance in low vision? A review of the literature. *Ophthalmic and Physiological Optics*. 2002;22(1):68-77.
- 3. Hickcox KS, Narendran N, Bullough JD, Freyssinier JP. Effect of different coloured luminous surrounds on LED discomfort glare perception. *Lighting Research and Technology*. 2013;1477153512474450.

- 4. Leguire LE, Suh S. Effect of light filters on contrast sensitivity function in normal and retinal degeneration subjects. *Ophthalmic and Physiological Optics*. 1993;13(2):124-128.
- 5. Morse RS. Glare filter preference: influence of subjective and objective indices of glare, sharpness, brightness, contrast and color. *In Proceedings of the Human Factors and Ergonomics Society Annual Meeting*. 1985;Vol. 29, No. 8, pp. 782-786. SAGE Publications.
- 6. Pérez-Carrasco MJ, Puell MC, Sánchez-Ramos C, López-Castro A, Langa A. Effect of a yellow filter on contrast sensitivity and disability glare after laser in situ keratomileusis under mesopic and photopic conditions. *Journal of Refractive Surgery*. 2005;21(2):158-165.
- 7. Sheedy JE, Hayes J, Engle J. Is all asthenopia the same? *Optometry & Vision Science*. 2003;80(11):732-739.
- 8. Steen R, Whitaker D, Elliott DB, Wild JM. Age-related effects of glare on luminance and color contrast sensitivity. *Optometry & Vision Science*. 1994;71(12):792-796.
- 9. Vincent AJ, Spierings EL, Messinger HB. A controlled study of visual symptoms and eye strain factors in chronic headache. *Headache: The Journal of Head and Face Pain*. 1989;29(8):523-527.
- 10. Wilkins AJ, Evans BJ. Visual stress, its treatment with spectral filters, and its relationship to visually induced motion sickness. *Applied Ergonomics*. 2010;41(4):509-515.

## 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

# 2.1. Objectives

## Primary Objective

The primary objective of this study is to demonstrate non-inferiority of the Test lens compared to the Control lens with respect to CLUE comfort, Slit Lamp Findings (Grade 3 or Higher) and Distance Monocular logMAR Visual Acuity. This study will also aim to show that the Fit Acceptance rate is at least 90% while wearing the Test lens.

## Secondary Objective

The secondary objective of this study is to demonstrate non-inferiority of the Test lens compare to the Control lens with respect to CLUE Overall quality of Vision and Handling.

# **Exploratory Objective**

This study also aims to explore the performance of Indoor, Outdoor and Driving performance using individual questionnaire items.

## 2.2. Endpoints

Primary Endpoints
Primary Efficacy Endpoints:

## **CLUE Overall Comfort**

Overall comfort scores will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>)<sup>5</sup> questionnaire at the two-week follow-up. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.

## Distance Monocular Contact Lens Visual Acuity

Distance monocular contact lens visual performance (logMAR) is assessed for each subject eye at the two-week follow-up evaluation using EDTRS charts under two lighting conditions, (1) Bright illumination low contrast and (2) Dim Illumination High Contrast.

# Vision Satisfaction in Bright Lighting

Vision satisfaction in bright lighting will be assessed using the individual item (Item ID: V015\_1) "I was satisfied with the quality of my vision in bright lighting" from the CLUE<sup>TM</sup> questionnaire. This item uses the response scale, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree.

Primary Safety Endpoints:

## Slit Lamp Findings (Grade 3 or Higher)

Slit Lamp Findings will be assessed for each subject eye at all study visits (schedule and unscheduled). The percentage of eyes with Grade 3 or higher slit lamp findings will be analyzed and will include corneal infiltrates.

# Fit Acceptance Rate

Acceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each subject eye. Fit acceptance rate will be based on the lens fit acceptance of eyes wearing the Test lens only. Fit rates of the Control lens will also be collected but are not a primary endpoint.

# Secondary Endpoints

# CLUE Overall Quality of Vision and Handling

Overall Quality of vision and handling scores will be assessed using the Contact Lens User Experience (CLUE)<sup>5</sup> questionnaire at the two-week follow-up.

# Overall Quality of Vision Outdoors

Overall quality of vision outdoors will be assessed using the individual item (Item ID: MIS00622) "Overall quality of vision outdoors" from the market research questionnaire. This item uses the response scale, 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor.

#### Other Observations

# Lens Preferences

Lens preferences will be assessed by patient reported outcome (PRO) questions regarding lens preference at the two-week follow-up of the second wearing period (Visit 3). Subjects will be asked to choose for each preference item one of the following responses: Strongly Prefer the first lens, Prefer the first lens, no preference, prefer the second lens, strongly prefer the second lens. Lens preference questions consist of:

Overall lens preference
 Overall comfort
 Overall vision
 Overall reduction of glare
 Overall preference indoors
 Overall preference outdoors
 Overall preference while driving during the day
 Overall preference while driving at night
 Overall preference while using computer screens & digital devices

# **Driving Performance**

Driving performance will be assessed by two individual patient reported outcome (PRO) questions at the two-week follow-up evaluation. The individual items are as follows:

Reduction in glare while driving during the day
 Reduction in glare while driving during the night

#### **Indoor Performance**

Indoor performance will be assessed by three individual patient reported outcome (PRO) questions at the two-week follow-up evaluation. The individual items are as follows:

Reduction in glare from the computer screen or digital devices
 Reduction in glare caused by bright indoor lights
 Reduction in glare caused by bright light coming through the window

# **Outdoor Performance**

Outdoor performance will be assessed by four individual patient reported outcome (PRO) questions at the two-week follow-up evaluation. The individual items are as follows:

Ability to see comfortably in bright sunlight
 Reduction in glare in bright sunlight
 Reduction in squinting in bright sunlight
 Reduction in eye strain in bright sunlight

All driving, indoor and outdoor (PRO) items above will be assessed using the same excellence scale of; 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor.

Quick Contrast Sensitivity will also be evaluated during this study.

# 2.3. Hypotheses

# Primary Hypotheses

All primary and secondary hypotheses must be met to satisfy the objective the study.

| Primary Hypotheses | |
|---|---|
| Endpoint | Hypothesis |
| Monocular logMAR visual acuity | The Test lens will be non-inferior to the Control lens with respect to Distance Monocular logMAR Visual Acuity at the two-week follow-up evaluation under both lighting conditions (Bright illumination low contrast and dim illumination high contrast). A non-inferiority margin of 0.05 logMAR will be used. |
| Biomicroscopy | The Test lens will be non-inferior to the Control lens with respect to the percentage of eyes with Grade 3 or higher Slit Lamp Findings (Biomicroscopy) across all follow-up visits (scheduled and unscheduled). A non-inferiority odds ratio margin of 2 will be used. |
| Fit acceptance rate | The proportion of eyes with acceptable fit will be greater than 90% across all visits (scheduled and unscheduled) for all subjects wearing the Test lens. |
| Overall CLUE comfort | The Test lens will be non-inferior to the Control lens with respect to CLUE Overall Comfort at the two-week follow-up evaluation. A non-inferiority margin of -5 points will be used |
| Vision Satisfaction in<br>Bright Lighting | The Test lens will be non-inferior to the Control lens with respect to Vision satisfaction in bright lighting at the two-week follow-up evaluation. A non-inferiority cumulative odds ratio margin of 0.67 will be used. |

# Secondary Hypotheses

| Secondary Hypotheses | |
|---|---|
| Endpoint | Hypothesis |
| Overall CLUE Vision | The Test lens will be non-inferior to the Control lens with respect to CLUE Overall quality of vision at the two-week follow-up evaluation. A non-inferiority margin of -5 points will be used. |
| Overall CLUE handling | The Test lens will be non-inferior to the Control with respect to CLUE Handling at the two-week follow-up evaluation. A non-inferiority margin of -5 points will be used. |
| Overall Quality of<br>Vision Indoors | The Test lens will be non-inferior the Control lens with respect to Overall quality of vision indoors at the 2-week follow-up evaluation. A non-inferiority cumulative odds ratio margin of 0.67 will be used. |

# Other Hypotheses

| Other Observations | |
|---|---|
| Endpoint | Hypothesis |
| Lens Preferences | The Test lens will be superior to the Control lens in all 9 of the following lens preference items at the two-week follow-up evaluation of the second wearing period. 1. Overall lens preference 2. Overall comfort 3. Overall vision 4. Overall reduction of glare 5. Overall preference indoors 6. Overall preference outdoors 7. Overall preference while driving during the day |
| | <ul> <li>8. Overall preference while driving at night</li> <li>9. Overall preference while using computer screens &amp; digital devices</li> </ul> |

| Other Observations | |
|---|---|
| Endpoint | Hypothesis |
| | The Test lens will be superior to the Control lens in at least 2 of the following 4 indoor performance measure(s) at the two-week follow-up evaluation. |
| Indoor Performance<br>Measures | <ol> <li>Reduction in squinting while using computer screens or digital devices</li> <li>Reduction in glare from the computer screen or digital devices</li> <li>Reduction in glare caused by bright indoor lights</li> <li>Reduction in glare caused by bright light coming through the window</li> </ol> |
| Driving Performance<br>Metrics | The Test lens will be non-inferior to the Control lens with respect to both of the following driving performance metrics at the two-week follow-up evaluation. A cumulative odds ratio margin of 0.67 will be used. 1. Reduction in glare while driving during the day 2. Reduction in glare while driving during the night |
| Outdoor Performance | The Test lens will be superior to the Control lens in at least 2 of the following 4 outdoor performance measure(s) at the two-week follow-up evaluation. |
| Measures | <ol> <li>Ability to see comfortably in bright sunlight</li> <li>Reduction in glare in bright sunlight</li> <li>Reduction in squinting in bright sunlight</li> <li>Reduction in eye strain in bright sunlight</li> </ol> |
| Quick Contrast<br>Sensitivity | At the 2-week follow-up evaluation, the difference in the area under the contrast sensitivity function curve (measured by the quick Contrast Sensitivity Function (qCSF) method) between the Test lens and the Control lens is more than -0.3 log unit. |

# 3. TARGETED STUDY POPULATION

## 3.1. General Characteristics

Approximately 120 subjects will be enrolled to ensure that at least 105 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 and ≤49 years old. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear the Test and Control contact lenses approximately 2 weeks each bilaterally on a DW basis, then wear either the Test or Control lens again for 2 weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

# Inclusion Criteria after Screening

- 1. The subject must read and sign the Informed Consent form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Healthy adult males or females age ≥18 and ≤49 years of age with signed informed consent.
- 4. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them
- 5. Subjects must own a wearable pair of spectacles.
- 6. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis
- 7. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week
- 8. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

## Inclusion Criteria after Baseline

- 9. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and -6.00 D.
- 10. The subject's refractive cylinder must be  $\leq$ -1.00 D in each eye.
- 11. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

## Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
- 2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic

- Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
- 4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
- 5. Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multipurpose care solution or Eye-Cept® rewetting drop solution.
- 6. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 7. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 8. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
- 9. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).
- 10. Toric, extended wear, monovision or multi-focal contact lens correction.
- 11. History of binocular vision abnormality or strabismus.

## Exclusion Criteria after Baseline

- 12. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g.., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
- 13. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
- 14. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.

## 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

## 4. STUDY DESIGN AND RATIONALE

## 4.1. Description of Study Design

This study is a randomized, 4-visit, partially subject-masked, 2x3 bilateral crossover, dispensing trial. Approximately 120 subjects will be screened and enrolled to ensure that at least 105 subjects to complete.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, they will be randomized to one of two lens wear sequences (Test/Control/Control or Control/Test/Test).

If the subject is dispensed study lenses at the initial visit, 3 follow-up visits will be conducted. The follow-up visits occur approximately 2, 4 and 6 weeks after the initial visit. Unscheduled follow-up visits may occur during the study. Subjects will be advised to wear the study lenses at least five (5) days per week for at least six (6) hours per day for a period of two weeks each. Lens replacement is scheduled at 2 and 4-week follow-up visits.

## 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. This design was considered since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared a parallel study since fewer subjects are required to achieve the same pre-specified statistical power. In previous studies involving the Test lens clinically relevant differences between the Test lens and a comparator while using a 2×2 crossover study design. Therefore, a higher order 2x3 crossover will be utilized since in this design we are able to obtain within-subject estimators of the carryover effect and the direct-by-period interaction of these effects are not aliased with each other.

## 4.3. Enrollment Target and Study Duration

Approximately 120 subjects will be enrolled to ensure that at least 105 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 and  $\leq$ 49 years old. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear the Test and Control contact lenses bilaterally approximately 2 weeks each on a DW basis, then wear either the Test or Control lens again for 2 weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

# 5. TEST ARTICLE ALLOCATION AND MASKING

#### **5.1. Test Article Allocation**

Using a computer-generated randomization scheme will be used to randomly assign subjects, in blocks of 2, to one of the two possible lens wear sequences (TEST/CONTROL/CONTROL or CONTROL/TEST/TEST). The random scheme will be generated using the PROC PLAN procedure from SAS Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment according to the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected.

## 5.2. Masking

Complete masking is impossible due to the functioning nature of the Test lens. The Control lens will be over-labeled to mask the identity since the Control lens may be the subject's habitual lens by chance. Therefore, the study is partially-subject masked (Control lens only).

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may in an emergency contact the medical monitor. In the event the mask is broken, the sponsor must be notified before the mask is broken. The date, time, and reason for the unmasking must be documented in the source document. The investigator is also advised not to reveal the study treatment assignment to the study site or sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

If the test article is randomized, the order will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

# 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

## 6. STUDY INTERVENTION

## 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| ruble 1. Test Thireles | | |
|---|---|---|
| | Control | Test |
| Name | OASYS | ECL100 |
| Manufacturer | JJVC | JJVC |
| | | pr. |
| Lens Material | senofilcon A | senofilcon A |
| Nominal Base Curve @ 22°C | 8.4 | 8.4 |
| Nominal Diameter @ 22°C | 14.0 | 14.0 |
| Nominal Distance Powers (D) | -1.00 to -6.00 in | -1.00 to -6.00 in |
| | 0.25 steps | 0.25 steps |
| Water Content (Optional) | 38 | 38 |
| Center Thickness (Optional) | 0.070 | 0.085 |
| Oxygen Permeability (Dk) | 103 | 103 |
| Modality in Current Study | Daily wear | Daily wear |
| Replacement Frequency | Single use | Single use |
| Packaging Form (vial, blister, etc.) | Sterile blister pack | Sterile blister pack |
| New-UV blocker concentration | NA | ~1.0% |

Approximately 75 lenses per sku will be made available based on the following factors: sample size, 2×3 design, bilateral wear, biweekly replacement, safety margin of 2x, and US distribution model for the range of lenses -1.00 through -6.00 D.

# 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution 1 | Solution 2 |
|---|---|---|
| Solution Name /<br>Description | Opti-Free® PureMoist® | Eye-Cept®<br>Rewetting Drops |
| Lot Number or Other Identifier | Varies | Varies |
| Manufacturer | Alcon Laboratories, Fort Worth, TX | Optics<br>Laboratories |
| Maximum<br>Preservative | 0.001% polyquaternium-1, 0.0006% myristamidopropyl dimethylamine | NA |

## 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an

adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

# 6.4. Packaging and Labeling

The Test articles will be packaged in blisters as the primary packaging. The Control article will be over-labeled to mask the subject to the identity of the lens. The Test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:

US label A (for Control lens over-label)

# **6.5. Storage Conditions**

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions and out of direct sunlight.

## 6.6. Collection and Storage of Samples

All worn study lenses will be collected from the subject, placed in labeled glass vials with Opti-Free® Puremoist®, and stored refrigerated or frozen until they are shipped back to the Sponsor. The lenses will be shipped in special containers to keep the lenses refrigerated.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

# 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will package and return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

# 7. STUDY EVALUATIONS

# 7.1. Time and Event Schedule

Table 3: Time and Events

| Procedure | Baseline | Trial Fit & Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 2, 3 | 2, 3, 4 | PRN | 4 |
| Visit Window | - | - | 13-15 Days | - | - |
| Estimated Visit Duration | - | V1: 2 hours | V2, 3: 1 hour<br>V4: 1.5 hours | - | - |
| Informed consent | ✓ | - | - | - | - |
| Eligibility screening | ✓ | - | - | - | - |
| CLUE Baseline Questionnaire | ✓ | - | - | - | - |
| GSI Background Questionnaire | <b>√</b> | | | | |
| Other Questionnaires | ✓ | - | ✓ | - | - |
| Subject demographics | <b>√</b> | - | - | - | - |
| General health and medication history | <b>√</b> | - | - | - | - |
| Subject's own contact lens information | <b>√</b> | - | - | - | - |
| Habitual lens care | <b>√</b> | - | - | - | - |
| Entrance visual acuity | <b>√</b> | - | - | - | - |
| Spherocylindrical refraction and BVA | <b>√</b> | - | - | <b>√</b> | <b>√</b> |
| Slit lamp biomicroscopy | <b>√</b> | - | ✓ | ✓ | - |
| Expanded Conjunctival<br>Redness | ✓ | - | ✓ | <b>√</b> | - |
| Expanded Corneal Staining | <b>√</b> | - | <b>√</b> | <b>√</b> | - |
| Trial fitting lens information | _ | ✓ | - | - | - |
| Lens Damage | _ | ✓ | - | - | _ |
| Distance spherical over-<br>refraction | - | <b>√</b> | ✓ | - | - |
| Lens modification | _ | <b>√</b> | _ | _ | _ |
| Visual acuity | _ | <b>√</b> | <b>√</b> | <b>√</b> | _ |
| logMAR acuity | _ | _ | <b>√</b> | _ | _ |
| Contrast sensitivity (site 1036) | _ | _ | <b>√</b> | - | _ |
| Lens fitting assessment | _ | <b>√</b> | <b>√</b> | * | _ |
| Lens dispensing information and criteria | - | <b>√</b> | - | - | - |
| Patient instructions | - | <b>√</b> | - | - | - |
| Lens information | - | - | <b>√</b> | <b>√</b> | - |
| Compliance | _ | - | <b>√</b> | ✓ | - |
| Wearing times | _ | _ | ✓ | <b>√</b> | - |

| Procedure | Baseline | Trial Fit &<br>Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 2, 3 | 2, 3, 4 | PRN | 4 |
| Visit Window | , <del>, , </del> | | 13-15 Days | - | - |
| Estimated Visit Duration | ¥<br><b>E</b> 0 | V1: 2 hours | V2, 3: 1 hour<br>V4: 1.5 hours | ä | 8 <u>25</u> |
| CLUE Follow-Up<br>Questionnaire | ž | 8 | ✓ | * | |
| GSI Product Performance<br>Questionnaire | 悪り | ā. | ✓ | * | si <del>nt</del> s |
| Symptoms | , <del>, , </del> | <b>✓</b> | <b>√</b> | <b>√</b> | - |
| Lens preference | | :51 | V3 | = | 970 |
| Surface characteristics | 140 | <u>3</u> 28 | <b>√</b> | * | ~ |
| Chief complaint, diagnosis, treatment | æ0 | 5 | 8 <b>3</b> 7 | ✓ | g <del>irt</del> t |
| * if wearing study contact lens | es | 921 | , i | Į. | 10. |

# 7.2. Detailed Study Procedures

VISIT 1

Note that the subject must be wearing their habitual soft contact lenses into Visit 1.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Baseline<br>Questionnaires | The subject will respond to the following questionnaires: 1. CLUE Baseline Questionnaire 2. GSI Background Questionnaire |
| 1.7 | Other Questionnaires | The subject will respond to additional questionnaires: 1. Activity History |
| 1.8 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.9 | Remove Habitual<br>Lens | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. |
| 1.10 | Slit Lamp Findings | FDA Slit Lamp Classification Scale will be used to grade the findings and will be used to determine eligibility. Record only whole numbers. If any of these slit lamp findings are Grade 3 or higher, the subject is ineligible to continue but may return at a later date to complete another Baseline. If after a total of 2 attempts the subject is deemed ineligible, then complete the Final Evaluation. Limbal and Bulbar Conjunctival Hyperemia findings using the 0.5 increment scale, and Corneal Staining Assessment |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | will be emphasized using the 1.0 increment scale for internal purposes only. | |
| 1.11 | Iris Color | The investigator will record the subject's iris color based on the scale provided. | Appendix<br>E |
| 1.12 | Subjective<br>Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. Best corrected distance visual acuity (BVA) must be 20/25+3 or better in each eye. | |
| 1.13 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. | |
| 1.14 | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.15 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective refraction. |
| 1.16 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 1.17 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.18 | Spherical Over<br>Refraction and<br>Modification | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of $\pm 0.00$ D OD and OS. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | Ensure that any new lenses are not damaged. One modification attempt will be allowed. |
| 1.19 | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |
| 1.20 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.21 | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 1.22 | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 1.23 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Snellen visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 1.24 | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> </ol> |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | <ol> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>A patient instruction booklet will be provided.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> </ol> |
| | | Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit). |
| | | Note 2: The subject's habitual contact lenses cannot be worn at any time during the study. |
| | | Note 3: The subject must be instructed: At each of your follow-up visits in this research study, we'll ask about the lenses you're wearing. These questions will address lens comfort and vision, including color perception in different lighting conditions and the ability to see comfortably in bright light |

VISIT 2

The follow-up will occur 13-15 days following Visit 2. The subjects must enter the visit wearing their study contact lenses.

| | Visit 2: Treatment 1 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. |
| 2.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |

| Visit 2: Treatment 1 Follow-Up | | | |
|---|---|---|--|
| Step | Procedure | Details | |
| 2.5. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | |
| 2.6. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 2.7. | Quick Contrast<br>Sensitivity | only. Perform the 4 m contrast sensitivity test once OD and OS using the 25-item methodology while wearing the study lenses. | |
| 2.8. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS LogMAR visual acuity test OD and OS under the following conditions: 1. Bright room illumination / low contrast charts a. Room illumination >400 lux b. Chart luminance 120-200 cd/m² c. One low contrast chart per eye. 1) OD: chart LC-1 2) OS: chart LC-2 2. Low room illumination / high contrast charts a. Room illumination <2.5 lux b. Chart luminance 2.0-5.0 cd/m² c. One high contrast chart per eye. 1) OD: chart HC-1 2) OS: chart HC-1 2) OS: chart HC-2 | |
| 2.9. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories | |
| | Visit 2: Treatment 1 Follow-Up | | | |
|---|---|---|--|--|
| Step | Procedure | Details | | |
| 2.10. | Surface Deposits | Record any front and back surface lens deposits. | | |
| 2.11. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free <sup>®</sup> PureMoist <sup>®</sup> . The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVC for 45 days after LSLV for laboratory testing (Section 7.4). | | |
| 2.12. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be grade 2 or less as graded on the FDA scale continue onto Trial Period 2. If the subject is not eligible, they must be followed as an | | |
| | | adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. | | |
| 2.13. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. | | |

| | Visit 2: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 2.14. | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective refraction or the final lens power from Period 1. |
| 2.15. | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. |

| | Visit 2: Treatment 2 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Check for lens damage under the slit lamp<br>before proceeding with lens settling.<br>Replace damaged lenses if applicable. | |
| 2.16. | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. | |
| 2.17. | Spherical Over<br>Refraction and<br>Modification | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. | |
| 2.18. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. | |
| 2.19. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 2.20. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. | 3e − |

| Visit 2: Treatment 2 Lens Fitting | | |
|---|---|---|
| Step | Procedure | Details |
| 2.21. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |

| | Visit 2: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 2.22. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 2.23. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> </ol> |

# VISIT 3

The follow-up will occur 13-15 days after the dispensing of the second study lenses. The subjects must enter the visit wearing their study contact lenses.

| Visit 3: Treatment 2 Follow-Up | | |
|---|---|---|
| Step | Procedure | Details |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. |

| | Visit 3: Treatment 2 Follow-Up | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Record any adverse events or medical history changes from the previous study visit. | |
| 3.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | 11 |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. | |
| 3.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.5. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | |
| 3.6. | Lens Preferences | Subjects will respond to the preference questionnaire comparing study lens 1 and study lens 2. | |
| 3.7. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | 7.6 |
| 3.8. | Quick Contrast<br>Sensitivity | Site 1036 only. Perform the 4 m contrast sensitivity test once OD and OS using the 25-item methodology while wearing the study lenses. | |
| 3.9. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS LogMAR visual acuity test OD and OS under the following conditions: 1. Bright room illumination / low contrast charts a. Room illumination >400 lux b. Chart luminance 120-200 cd/m² c. One low contrast chart per eye. 1) OD: chart LC-1 2) OS: chart LC-2 2. Low room illumination / high contrast charts a. Room illumination <2.5 lux | |

| | Visit 3: Treatment 2 Follow-Up | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | <ul> <li>b. Chart luminance 2.0-5.0 cd/m²</li> <li>c. One high contrast chart per eye.</li> <li>1) OD: chart HC-1</li> <li>2) OS: chart HC-2</li> </ul> | |
| 3.10. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift Insufficient and/or excessive movement in all three movement categories | |
| 3.11. | Surface Deposits | Record any front and back surface lens deposits. | 5.0 |
| 3.12. | Lens Removal & Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). | |
| 3.13. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be grade 2 or less as graded on the FDA scale continue onto Trial Period 2. If the subject is not eligible, they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. | |
| 3.14. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. | |

| | Visit 3: Treatment 3 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.15. | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective refraction or from Period 2 final lens power. Record the test condition. | |
| 3.16. | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. | |
| 3.17. | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. | |
| 3.18. | Spherical Over<br>Refraction and<br>Modification | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. | |
| 3.19. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. | 35 |
| 3.20. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.21. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. | |
| 3.22. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift | |

| | Visit 3: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | Insufficient and/or excessive movement in all three movement categories |
| 3.23. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 3.24. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> </ol> |

# VISIT 4 The follow-up will occur 13-15 days after the dispensing of the third study lenses. The subjects must enter the visit wearing their study contact lenses.

| | Visit 4: Treatment 3 Follow-Up | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. | |
| 4.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. | |
| 4.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 4.5. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | 4.0 |
| 4.6. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 4.7. | Quick Contrast<br>Sensitivity | Site 1036 only. Perform the 4 m contrast sensitivity test once OD and OS using the 25-item methodology while wearing the study lenses. | |

| | Visit 4: Treatment 3 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| 4.8. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS LogMAR visual acuity test OD and OS under the following conditions: 1. Bright room illumination / low contrast charts a. Room illumination >400 lux b. Chart luminance 120-200 cd/m² c. One low contrast chart per eye. 1) OD: chart LC-1 2) OS: chart LC-2 2. Low room illumination / high contrast charts a. Room illumination <2.5 lux b. Chart luminance 2.0-5.0 cd/m² c. One high contrast chart per eye. 1) OD: chart HC-1 2) OS: chart HC-1 2) OS: chart HC-2 |
| 4.9. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 4.10. | Surface Deposits | Record any front and back surface lens deposits. |
| 4.11. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). |

| | Visit 4: Treatment 3 Follow-Up | |
|---|---|---|
| Step | Step Procedure Details | |
| 4.12. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be Grade 2 or less as graded on the FDA scale Otherwise they must be followed as an adverse event. Adverse events must be reported to the JJVC monitors immediately. |
| 4.13. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| Final Evaluation | | |
|---|---|---|
| Step | Step Procedure Details | |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |
| F.2 | Best-corrected Distance<br>Visual Acuity | Record the subject's best corrected distance visual acuity with refraction OD, OS, and OU. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Step | Procedure | Details |
|---|---|---|
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Change of Medical<br>History and Concomitant<br>Medications | Questions regarding the change of subjects' medical history and concomitant medications. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.4 | Subjective Sphero-<br>cylindrical Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. |
| U.5 | Slit Lamp Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If no slit lamp finding is noted on the EDC form it is considered as a zero "0" Grade for all observations listed. After the slit lamp examination, at the discretion of the Investigator, rinse the subject's eyes thoroughly with preservative-free saline. |
| U.6 | Dispensing (if applicable) | Additional lenses may be dispensed if one is lost or torn during the wearing period. |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS and OU) to the nearest letter. |

## 7.4. Laboratory Procedures

The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- completed all scheduled visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol (e.g. Subject more than 2 days out of visit window).
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear (subjects missing more than 2 days of missed lens wear within a period 1 of week should be discontinued)
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed any scheduled study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2.
- Collect all unused test article(s) from the subject

Investigator will discuss with sponsor before enrolling any additional subjects if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to

follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: See Section 3.3 Concomitant therapies that are disallowed include: See Section 3.3

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)".
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13of this

protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

**Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions

• Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; doubtful; possible; probable; very likely see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2).
- Outcome not Recovered or Not Resolved; Recovering or Resolving; Recovered or Resolved with Sequelae; Recovered or Resolved; Death Related to Adverse Event; Unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

#### 13.2.1 Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant

- treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

## 13.2.2 Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution

- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment /eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the test article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1 Reporting Adverse Events to Sponsor

# **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24

hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.4.3 Event of Special Interest

None.

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

This section is a general outline of the statistical methods that will be implemented in this clinical trial. More details will be included in the stand-alone Statistical Analysis Plan (SAP). The SAP will be developed and finalized prior to database lock.

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

This study was designed and powered to show non-inferiority of the Test lens compared to the Control lens with respect to logMAR Visual Acuity, Slit Lamp Findings (Grade 3 or higher), CLUE comfort, handling and overall quality of vision. It was assumed there was no difference between the Test and Control lens with respect to visual acuity and slit lamp findings. Based on data from 3 historical studies, it was assumed there was a 5-, 3- and 4-point difference between the Test and Control lenses with respect to CLUE comfort, handling and overall quality of vision, respectively.

In addition to the endpoints mentioned above this study was also powered to demonstrate non-inferiority of the Test lens relative to the Control lens with respect to vision satisfaction in

bright lighting, overall quality of vision indoors and the proportion of eyes with acceptable fitting while the Test lens is significantly superior to 90%.

Unless otherwise specified, the sample size was calculated to achieve a minimum statistical power of 80% and a type I error of 5%.

A total of 5 historical studies were utilized in the sample size calculation. Table 4 displays the studies, their corresponding study design and the number of subjects enrolled and completed per-protocol.

Table 4: Historical Studies Included in Sample Size Calculation

| Study | Study Design | <b>Endpoints Collected</b> | No.<br>Enrolled | No. Completed<br>Per-Protocol |
|---|---|---|---|---|
| | 2X3 Crossover | CLUE, SLF Lens Fit | 135 | 132 |
| | 2X3 Crossover | CLUE, Visual Acuity (logMAR), SLF, Lens Fit | 133 | 121 |
| | 2X3 Crossover | CLUE, SLF Lens Fit | 92 | 78 |
| | Single-Arm | SLF, Lens Fit | 54 | 48 |
| | Single-Arm | SLF, Lens Fit | 56 | 41 |

Table 5: Descriptive Summary of CLUE Scores by Domain Pooled Across Historical Studies

| | – 2-Week Follow-up Evaluation | |
|---|---|---|
| CLUE Domain [Mean(SD) <sup>1</sup> ] | Test | Control |
| Comfort | 66.46 (22.20) | 61.19 (24.20) |
| Handling | 69.61 (19.18) | 66.79 (20.01) |
| Overall Quality of Vision | 64.15 (18.83) | 60.33 (22.29) |

<sup>1</sup>SD = Standard Deviation

Evaluation

| Visual Acuity High<br>Illumination High | | |
|---|---|---|
| Contrast | Test | Control |
| [Mean(SD) <sup>1</sup> ] | -0.0928 (0.08253) | -0.0726 (0.08011) |

<sup>&</sup>lt;sup>1</sup>SD = Standard Deviation

Table 7: Descriptive Summary of Mechanical Lens Fitting Pooled Across all Historical Studies

| Any Unacceptable Lens Fit <sup>1</sup> [n(%)] | Test n (%) | Control n (%) |
|-----------------------------------------------|------------|---------------|
| Fitting Evaluation | 0(0.0) | 0 (0.0) |
| 2-Week Follow-up | 0 (0.0) | 0 (0.0) |

<sup>&</sup>lt;sup>1</sup>The percent of any unacceptable fit is calculated using Total Unique eyes as a denominator

Table 8: Descriptive Summary of Slit Lamp Findings Pooled Across all Historical Studies

| SLF Grade 2 | Test n (%) | Control n (%) |
|------------------------------|-------------|---------------|
| Corneal Edema | 0 (0.0) | 0 (0.0) |
| Conjunctival Injection | 59 (6.86) | 59 (21.85) |
| Tarsal Abnormalities | 51 (5.93) | 24 (8.89) |
| Corneal Neovascularization | 3 (0.35) | 0 (0.0) |
| Corneal Staining | 3 (0.35) | 0 (0.0) |
| Other Findings | 0 (0.0) | 0 (0.0) |
| Total Eyes (N) | 860 | 270 |
| Any SLF Grade 2 <sup>2</sup> | 116 (13.48) | 83 (33.74) |
| Any SLF Grade 3+ | 0 (0.0) | 0 (0.0) |
| Total Unique Eyes | 860 | 270 |
| Total Unique Subjects | 430 | 135 |

<sup>%=</sup> nx100/N; SD=Standard Deviation

<sup>&</sup>lt;sup>1</sup>All SLF reported for this study are combined for the purposes of summarizing

<sup>&</sup>lt;sup>2</sup> The percent (%) of Any Grade 2 is calculated using the Total Unique Eyes as the denominator

| Гable 9: Descriptive Summary of Individu | al Items from $-2$ -V | Week Follow-up |
|---|---|---|
| Questionnaire Item/ Response | Test | Control |
| Vision Satisfaction in Bright Light [n(% | <b>6</b> )] | |
| Strongly Agree | 72 (29.75) | 51 (21.07) |
| Agree | 129 (53.31) | 130 (53.72) |
| Neither Agree Nor Disagree | 24 (9.92) | 21 (8.68) |
| Disagree | 17 (7.02) | 33 (13.64) |
| Strongly Disagree | 0 (0.0) | 7 (2.89) |
| Overall Quality of Vision Indoors [n (% | <b>%</b> )] | |
| Excellent | 100 (55.25) | 80 (43.96) |
| Very Good | 55 (30.39) | 62 (34.07) |
| Good | 23 (12.71) | 30 (16.48) |
| Fair | 3 (1.66) | 7 (3.85) |
| Poor | 0 (0.0) | 3 (1.65) |

# **CLUE Comfort**

Sample size calculation for CLUE comfort was carried out using an approximation of the power of an F-test derived from the non-centrality parameter calculated form the observed F statistic of a linear model<sup>12</sup>.

#### Model details:

CLUE comfort was analyzed using a linear mixed model. Lens type was included as the only fixed effect. An unstructured (UN) covariance matrix was used to model the correlation between measurements on the same subject across study periods. Below is the variance-covariance matrix used in the CLUE Comfort model.

$$\sum_{comfort} \begin{pmatrix} 397.18 & 142.48 & 144.55 \\ 142.48 & 411.89 & 210.90 \\ 144.55 & 210.90 & 370.83 \end{pmatrix}$$

## **Visual Performance (logMAR)**

Sample size calculation for visual performance (logMAR) was carried out using an approximation of the power of an F-test derived from the non-centrality parameter calculated form the observed F statistic of a linear model<sup>12</sup>.

#### Model details:

visual performance was analyzed using a linear mixed model. Lens type was included as the only fixed effect. A compound symmetric (CS) covariance matrix was used to model the correlation between measurements on the same subject across study periods. Below is the variance-covariance matrix used in the visual performance model.

$$\sum_{visual\ performance} \begin{pmatrix} 0.003518 & 0.000374 & 0.000374 \\ 0.000374 & 0.003518 & 0.000374 \\ 0.000374 & 0.000374 & 0.003518 \end{pmatrix}$$

## **Acceptable Lens Fit**

Acceptable lens fit is a binary response as y=1 if a subject eye has an acceptable fit and 0 otherwise. Indicated by the historical data there were no observed unacceptable lens fittings for either the Test or Control lens therefore, the common reference rate of 95% was selected for the sample size calculation, since this is considered to be a more conservative reference proportion. Assuming a correlation 0.80 between measurements within the same subject and period; and assuming a correlation of 0.50 between measurements within the same subject across periods. A total of 2000 replicating trials were simulated to estimate a sample size with a minimum statistical power of 80%.

## **Slit Lamp Findings**

There were no Grade 3 or higher SLFs observed in any of the historical studies. Assuming no difference between study lenses and a correlation 0.80 between left and right eyes within the same subject and period; and a correlation of 0.50 between measurements within the same subject across periods (intra-subject correlation). A reference rate of no more than 10% was assumed (worse-case scenario) with a non-inferiority odds ratio margin of 2. A total of 2000 replicating trials were simulated, each replicated sample was analyzed using a generalized estimating equation (GEE) model with a binary distribution and the logit as the link function. Each model included lens type as the only fixed, eye was included as a random effect. The Odds ratio and corresponding 95% confidence interval was used estimate differences between the Test and Control lenses. The upper limit of each 95% confidence interval was compared to 2; if the upper limit was below 2 then NI=1; otherwise NI=0. Statistical power was calculated at the average NI. A sample size of 50 was chosen to achieve a minimum statistical power of 80%.

The non-inferiority odds ratio margin of 2 corresponds to no more than a 5% difference between the Test and Control lenses assuming the Control reference rate does not exceed 10%.

#### **Individual Ouestionnaire Items**

Overall quality of vision outdoors and vision satisfaction in bright lighting sample size estimates were calculated using historical data from . One-thousand boot strap

samples were simulated based on the historical data. For each replicated sample a generalized linear mixed model was used with a multinomial distribution and the cumulative logit as the link function. Lens wear sequence, lens type, period and first order carryover effect were included in the model as fixed effects. A variance component (VC) covariance structure was used to model the measurements between subjects across study periods.

The non-inferiority cumulative odds ratio margin of 0.67 corresponds to no more than a 10% difference between the Test and Control lenses assuming there is no difference between study lenses.

Table 10: Sample Size Estimates and Power Calculations for Primary Endpoints

| Endpoint | Number per<br>Subjects to<br>Complete | Power |
|---|---|---|
| Distance Monocular Visual Acuity (logMAR) | 4 | 80% |
| SLFs (Grade 3 or Higher) | 50 | 80% |
| Acceptable lens Fit | 65 | 80% |
| CLUE Comfort | 30 | 87% |
| Vision Satisfaction in Bright Lighting | 48 | 81% |

Table 11: Sample Size Estimates and Power Calculations for Secondary Endpoints

| Endpoint | Number per Subjects to<br>Complete | Power |
|---|---|---|
| CLUE Handling | 30 | 81% |
| CLUE Overall Quality of Vision | 30 | 82% |
| Overall Quality of Vision Indoors | 95 | 81% |

As indicated in Table 10 and 11 above, the sample size chosen for this study was primary driven by overall quality of vision indoors. The plan is to enroll 120 eligible subjects with a target of 105 subjects to complete the study. During the enrollment period, the subject dropout rate with be closely monitored, if an unexpectedly high dropout rate is observed, then the targeted total enrollment number maybe be increased accordingly to ensure that a minimum of 105 subjects complete the study.

## 14.3. Analysis Populations

A separate SAP will be provided for this study. If there are any discrepancies between the protocol and the SAP, the SAP will supersede the statistical sections in the protocol.

## **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

The primary and secondary hypotheses will be tested with a type I error of 5% individually.

## 14.5. Primary Analysis

Primary efficacy analysis:

#### **Visual Acuity**

Distance monocular visual acuity (logMAR) will be tested under two conditions (bright illumination low contrast and dim illumination high contrast). Each condition will be analyzed separately using a Bayesian multivariate normal random-effects model to compare the Test and Control lenses. The regression model will include sequence of lens wear, lens type and first-order carryover effect as fixed effects. Clinical site and subject nested within clinical site will be included as random effects. Other subject characteristics such as gender and age will be included as fixed effects when appropriate.

## The Model:

Let  $y_{ijklm} = (y1_{ijklm}, y2_{ijklm}, y3_{ijklm})$  denote the visual acuity (logMAR) for the  $m^{th}$  subject at the  $l^{th}$  site, assigned to the  $i^{th}$  lens for the  $j^{th}$  eye using the  $k^{th}$  sequence at periods 1, 2, 3, respectively. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{ijklm} \sim N(\mu_{ijklm}, \Sigma)$$

Where  $\mu_{ijklm} = (\mu 1_{ijklm}, \mu 2_{ijklm}, \mu 3_{ijklm})^T$  and  $\Sigma$  is a 3X3 variance-covariance matrix. Here,

$$\mu 1_{ijklm} = \mu_0 + \pi_1 + \beta_1 Lens_{[i,k]} + \beta_2 Sequence_k + \gamma_l + \alpha_j$$

$$\mu 2_{ijklm} = \mu_0 + \pi_2 + \beta_1 Lens_{[i,k]} - \beta_2 Sequence_k + \beta_3 Carry 1_{[i,k]} + \gamma_l + \alpha_j$$

$$\mu 3_{ijklm} = \mu_0 + \pi_3 + \beta_1 Lens_{[i,k]} + \beta_2 Sequence_k - \beta_3 Carry 1_{[i,k]} + \gamma_l + \alpha_j$$

In this model  $\pi_1$ ,  $\pi_2$ ,  $\pi_3$  represent the effect of period with the constraint  $\pi_1 + \pi_2 + \pi_3 = 0$ . Lens will be determined by sequence k therefore lens i is denoted as a function of k. We define  $Lens_l = 0$  for the Control lens and  $Lens_i = 1$  for the Test lens, sequence is defined as: Sequence=0 for the order Control/Test/Test and Sequence=1 for order Test/Control/Control. The first-order carryover effect will be defined as carry=0 for the Control lens and carry=1 for the Test lens. So  $\beta_1$  stands for the difference between the Test and Control lens with respect to

visual performance at period 1. A negative  $\beta_1$  indicates the Test performed better than the Control lens.

We assume random subject eye effects are independent and identically distributed (i.i.d) as  $\alpha_j \sim N(0, \sigma_{eye}^2)$  as random eye and the random site effect is i.i.d as  $\gamma_l \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2 (sequence), carry1=1, 2 (first-order carryover effect) and l=1...|  $m_l$ (subject/site) and l=1,2,3,4,5 and 6 (site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effects  $\sigma_{eye}^2$  and  $\sigma_{site}^2$  independent non-informative conjugate priors inverse-gamma(0.001, 0.001) will be used. For  $\Sigma$ , non-informative conjugate priors inverse-wishart(3,S) will be used where S is a 3X3 variance-covariance matrix of  $y_{ijklm}$ . The metropolis sampler algorithm as implemented in the SAS/STAT MCMC 14.2<sup>14</sup> procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

## **Hypothesis Testing**

The null and alternative hypothesis for visual acuity (logMAR) to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o: \beta_1 \ge 0.05$$
  
 $H_A: \beta_1 < 0.05$ 

Non-inferiority will be declared if the upper limit of the 95% credible interval of the difference between the Test and Control is below 0.05, i.e.  $P(\beta_1 < 0.05) \ge 0.975$ .

## **CLUE Overall Comfort**

CLUE Comfort scores will be analyzed using a Bayesian multivariate normal random-effects model to compare the Test and Control lenses. The regression model will include baseline CLUE comfort scores, sequence of lens wear, lens type and first-order carryover effect as fixed effects. Clinical site will be included as random effects. Other subject characteristics such as age, gender, race and iris category will be included when appropriate.

## The Model:

Let  $y_{ijkl} = (y1_{ijkl}, y2_{ijkl}, y3_{ijkl})$  denote the CLUE Comfort score for the  $l^{th}$  subject at the  $k^{th}$  site, assigned to the  $i^{th}$  lens using the  $j^{th}$  sequence at periods 1, 2 and 3. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{ijkl} \sim N(\mu_{ijkl}, \Sigma)$$

Where 
$$\mu_{ijkl} = (\mu 1_{ijkl}, \mu 2_{ijkl}, \mu 3_{ijkl})^T$$
 and  $\Sigma$  is a 3X3 variance-covariance matrix. Here,  $\mu 1_{ijkl} = \mu_0 + \pi_1 + \beta_1 Lens_{[i,j]} + \beta_2 baseline + \beta_3 Sequence_j + \gamma_k$   $\mu 2_{ijkl} = \mu_0 + \pi_2 + \beta_1 Lens_{[i,j]} + \beta_2 baseline - \beta_3 Sequence_j + \beta_4 Carry 1_{[i,j]} + \gamma_k$   $\mu 3_{ijkl} = \mu_0 + \pi_3 + \beta_1 Lens_{[i,j]} + \beta_2 baseline + \beta_3 Sequence_j - \beta_4 Carry 1_{[i,j]} + \gamma_k$ 

In this model  $\pi_1$ ,  $\pi_2$ ,  $\pi_3$  represent the effect of period with the constraint  $\pi_1 + \pi_2 + \pi_3 = 0$ . Lens will be determined by sequence j, therefore i is denoted as a function of j. We define Lens=0 for the Control lens and Lens = 1 for the Test lens, sequence is defined as: Sequence=0 for the order Control/Test/Test and Sequence=1 for order Test/Control/Control. The first-order carryover effect will be defined as carry=0 for the Control lens and carry=1 for the Test lens. So  $\beta_1$  stands for the difference between the Test and Control lens at period 1 with respect to CLUE comfort; A positive  $\beta_1$  indicates the Test performed better than the Control.

We assume random site effects are independent and identically distributed (i.i.d) as  $\gamma_k \sim N(0, \sigma_{site}^2)$  for site for i=1, 2 (lens), j=1, 2 (sequence), k=1, 2, 3, 4, 5 and 6 (site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effect of  $\sigma_{site}^2$  an independent non-informative conjugate prior, inverse-gamma(0.001, 0.001) will be used. For  $\Sigma$ , non-informative conjugate priors inverse-wishart(3,S) will be used where S is a 3X3 variance-covariance matrix of  $y_{ijkl}$ . Starting values for the mean and variance of CLUE scores will be 60 and 400 (since standard deviation of CLUE is normalized to be 20), respectively. The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC 14.2<sup>14</sup> procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

## Hypothesis Testing

The null and alternative hypotheses for CLUE comfort non-inferiority of the Test lens relative to the Control lens are as follows:

$$H_o$$
:  $\beta_1 \leq -5$ 

$$H_A: \beta_1 > -5$$

Non-inferiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between the Test lens and the Control lens is greater than -5, i.e.,  $P(\beta_1 > -5) \ge 0.975$ .

## **Vision Satisfaction in Bright Lighting**

Vision satisfaction in bright lighting will be analyzed using a Bayesian multinomial model for ordinal data. The regression model will include sequence of lens wear, lens type, period and first order carryover effect. Clinical site and subject nested within clinical site will be included as random effects. Other subject characteristics such as age, gender, race and iris category will be included when appropriate.

#### The Model:

Let  $y_{ijklm} = (y_{ijklm1}, y_{ijklm2}, y_{ijklm3}, y_{ijklm4}, y_{ijklm5})$  denote the rating for the  $m^{th}$  subject, from the  $l^{th}$  site, assigned to the  $i^{th}$  study lens in the  $j^{th}$  period using the  $k^{th}$  sequence. Possible values of  $y_{ijklm}$  are 1 if the subject rating of vision satisfaction in bright lighting are X and 0 otherwise (x=1 for Strongly Agree and X=5 for Strongly Disagree, respectively). The likelihood is constructed as follows:

$$\begin{aligned} y_{ijklm} \sim \text{Multinomial} & (P_{ijklm1}, \ P_{ijklm2} \ , P_{ijklm3}, P_{ijklm4}, P_{ijklm5}) \\ & P_{ijklm1} = \gamma_{ijklm1} \\ & P_{ijklmX} = \gamma_{ijklmX} - \gamma_{ijklm(X-1)} \ 2 \leq n \leq 4 \\ & P_{ijklm5} = 1 - \sum_{x=1,..4} P_{ijklmX} \end{aligned}$$

$$\text{Logit(} \ \gamma_{ijklmX} \ ) = \ \theta_n \ + \ \beta_1 Lens_{i[j,k]} \ + \ \beta_2 Period_{j1} \ + \ \beta_3 Period_{j2} \ + \ \beta_4 Sequence_k \ + \ \beta_5 Carry_{i[j,k]} \ + \ \gamma_l + \delta_{m_{(l)}}$$

Where  $\theta_n$  is the intercept for levels n=1,2,3,4,  $P_{ijklm1} = \Pr(\gamma_{ijklm1} = 1)$  with respect to the vision satisfaction in bright lighting item. We assume the random subject effects are independent identically distributed (i.i.d) as  $\delta_{m_{(l)}} \sim N(0, \sigma_{subject}^2)$  for subject m nested within clinical site 1 and the random clinical site effects are i.i.d as  $\gamma_l \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2, 3 (Period) k=1, 2(Sequence) l=1, ...6 (Site) m=1, ... $n_l$ (subject/site).

In this model, the lens I will be determined by the period j and sequence k, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the Control lens and  $Lens_i=1$  for the Test lens. The odds ratio for having higher rating can be written as  $OR=e^{\beta 1}$ .

Independent vague N(0, 1000) priors for the regression coefficients  $\beta_i$  i=1,...5. For  $\theta_n$ , we are considering the following priors

$$\begin{array}{c} \pi 0(\theta 1) \sim N(0,100) \\ \pi 0(\theta 2|\: \theta 1) \sim N(0,100) I(\theta {>} \theta 1) \\ \pi 0(\theta 3|\: \theta 2) \sim N(0,100) I(\theta {>} \theta 2) \\ \pi 0(\theta 4|\: \theta 3) \sim N(0,100) I(\theta {>} \theta 3) \end{array}$$

For the variance of random effects independent vague normal priors will also be used;  $\sigma_P^2$  ~inverse-gamma(0.001, 0.001) and  $\sigma_s^2$  ~inverse-gamma(0.001, 0.001). The Metropolis sample algorithm as implemented in the SAS/Stat MCMC Procedure will be used to estimate the posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

## **Hypothesis Testing**

The null and alternative hypotheses for superiority are as follows:

$$H_o \ OR \le 0.67$$
  
 $H_A \ OR > 0.67$ 

Where OR represent the odds ratio of having higher rating of the Test lens compared to the Control lens. Non-inferiority will be declared if the lower bound of the 2-sided 95% credible confidence interval is above 0.67, i.e.  $P(OR=e^{\beta 1}>0.67|y)=0.975$ .

Primary Safety Analysis:

#### **Lens Fit Acceptance**

Lens fit acceptance will be analyzed using a Bayesian Logistic regression random-effects model to estimate the proportion of subjects' eyes wearing the Test lens having acceptable lens fitting. The regression model will include period, sequence of lens wear and first order carryover effect as fixed effects. Site, subject nested within site and eye within subject within site will be included in the model as random effects.

Let  $y_{ijklm}=1$  if an acceptable lens fit is observed for eyes wearing the Test lens only and  $y_{ijklm}=0$  otherwise for the  $m^{th}$  subject, from the  $l^{th}$  site, for the  $i^{th}$  eye in the  $j^{th}$  period using the  $k^{th}$  sequence.

$$y_{ijklm} \sim Binary (p_{ijklm})$$

$$p_{ijklm} = \frac{exp(\textit{Numerator})}{1 + exp(\textit{Numerator})}$$

$$\begin{aligned} Numerator &= \beta_0 + \beta_1 Lens_{i[j,k]} + \beta_3 period_{j1} + \beta_4 period_{j2} + \beta_5 sequence_k + \beta_6 Carry1_{i[j,k]} + \gamma_l + \delta_{m_{(l)}} + \alpha_{j_{(m(l))}} \end{aligned}$$

We assume the random subject eye effects are i.i.d as  $\alpha_{j_{(m(l))}} \sim N(0, \sigma_{eye}^2)$  for eye nested within subject within clinical site, the random effect for subject are i.i.d as  $\delta_{m_{(l)}} \sim N(0, \sigma_{subject}^2)$  for subject nested within clinical site and the random clinical site effects are i.i.d as  $\gamma_m \sim N(0, \sigma_{site}^2)$  for i=1, 2 (eye), j=1, 2, 3 (period) k=1, 2(Sequence) l=1, ...6 (Site) m=1, ... $n_l$ (subject/site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 10000) will be used. For the variance of random effects of  $\sigma_{eye}^2$ ,  $\sigma_{subject}^2$  and  $\sigma_{site}^2$ , independent non-informative conjugate priors inverse-gamma (0.001, 0.001) will be used. The Metropolis-Hastings algorithm as implemented in the SAS/STAT 14.2 PROC MCMC procedure will be used to estimate posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

## **Hypothesis Testing**

With respect to Acceptable lens fit the null and alternative hypothesis for superiority is as follows:

$$H_0 = p \le 0.90$$
  
 $H_1 = p > 0.90$ 

Where, p represents the proportion of subject eyes that achieve acceptable fit for the Test lens.

Success for acceptable fit will be declared if the lower bound of the 2-sided 95% credible interval of the proportion is greater than 0.90; i.e.  $P(P > 0.90) \ge .975$ .

If the full planned model fails to converge, reduced versions may be considered.

Primary safety analysis:

## **Slit Lamp Findings**

Grade 3 or higher slit lamp findings will be analyzed using a Bayesian Logistic regression random-effects model to compare the Test and Control lenses. The regression model will include baseline slit lamp findings, lens type, period, sequence of lens wear and first order carryover effect. Site, subject nested within site and eye within subject within site will be included in the model as random effects.

Let  $y_{ijklmn}$ =1 if a Grade 3 or higher SLF is observed and  $y_{ijklm}$  =0 otherwise for the  $n^{th}$  subject, from the  $m^{th}$  site, assigned to the  $i^{th}$  study lens for the  $j^{th}$  eye in the  $k^{th}$  period using the  $l^{th}$  sequence.

$$y_{ijklmn} \sim Binary\left(p_{ijklmn}\right)$$

$$p_{ijklmn} = \frac{exp(\textit{Numerator})}{1 + exp(\textit{Numerator})}$$

Numerator= 
$$\beta_0 + \beta_1 Lens_{ij[k,l]} + \beta_2 Baseline SLF_1 + \beta_3 period_{k1} + \beta_4 period_{k2} + \beta_5 sequence_k + \beta_6 Carry1_{i[k,l]} + \gamma_m + \delta_{n_{(m)}} + \alpha_{j_{(n(m))}}$$

We assume the random subject eye effects are i.i.d as  $\alpha_{j_{(n(m))}} \sim N(0, \sigma_{eye/subject/site}^2)$  for eye nested within subject within clinical site, the random effect for subject are i.i.d as  $\delta_{n_{(m)}} \sim N(0, \sigma_{subject/site}^2)$  for subject nested within clinical site and the random clinical site effects are i.i.d as  $\gamma_m \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2, 3 (period) l=1, 2 (Sequence) m=1, ...6 (Site) m=1, ... $n_m$  (subject/site).

In this model, the lens I will be determined by the period k and sequence l, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the Control lens and  $Lens_i=1$  for the Test lens. The odds ratio for having a lower rate of SLFs can be written as  $OR=e^{\beta 1}$ .

For the  $\beta$  coefficients, independent non-informative priors N(0, 10000) will be used. For the variance of random effects of  $\sigma_{eye}^2$ ,  $\sigma_{subject}^2$  and  $\sigma_{site}^2$ , independent non-informative conjugate priors inverse-gamma (0.001, 0.001) will be used. The Metropolis-Hastings algorithm as

implemented in the SAS/STAT 14.2 PROC MCMC procedure will be used to estimate posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

# **Hypothesis Testing**

The null and alternative hypothesis for Non-inferiority is as follows:

 $H_o$ : OR  $\geq 2$  $H_A$ : OR  $\leq 2$ 

Where OR represents the odds of the Test lens having a lower rate of Grade 3 SLFs compared to the Control lens. Non-inferiority will be established if the upper limit of the 2-sided 95% credible interval is below 2, i.e. P(OR < 2 | y) = 0.975.

If the full planned model fails to converge, reduced versions may be considered. In the event that the number of Grade 3 or higher SLFs is too small Grade 2 or higher SLFs will be analyzed and tested as described above.

# 14.6. Secondary Analysis

Secondary efficacy analysis:

## **CLUE Overall Quality of Vision and Handling**

CLUE Overall Quality of Vision and Handling will be analyzed and test in the exact same manner as CLUE Overall Comfort.

## **Overall Quality of Vision Indoors**

Overall quality of vision indoors will be analyzed and tested in the same manner as vision satisfaction in bright lighting. The only difference between the two models are the response set used to assess each item. For this model,

Let  $y_{ijklm} = (y_{ijklm1}, y_{ijklm2}, y_{ijklm3}, y_{ijklm4}, y_{ijklm5})$  denote the rating for the  $m^{th}$  subject, from the  $l^{th}$  site, assigned to the  $i^{th}$  study lens in the  $j^{th}$  period using the  $k^{th}$  sequence. Possible values of  $y_{ijklm}$  are 1 if the subject rating of overall quality of vision indoors are X and 0 otherwise (x=1 for Excellent and X=5 for Poor, respectively).

Secondary safety analysis:

Not Applicable

#### 14.7. Other Exploratory Analyses

Other efficacy analysis:

Lens preference, driving performance, indoor performance and outdoor performance will be descriptively summarized. Exploratory analysis on these items may be conducted.

Other safety analysis:

Not Applicable

## 14.8. Interim Analysis

An interim analysis will be conducted after the first 100 subjects complete the first wearing period or 4-weeks post first subject first visit. The interim analysis will consist of descriptively summarizing safety and efficacy parameters. The results will be reviewed with historical data with lenses from the pilot line before the design validation study, is initiated. The results will be communicated to study responsible clinician, project lead and platform lead.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 10 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Date Sources for this study include: If external Data is collected outside of EDC, enter vendor contact information in this section of the protocol and type of external data collected. Enter information for each external data source.

- Vendor Name:
- Vendor Address:
- Vendor Contact:
- Phone:
- Email:
- Type of Data collected:

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and

completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.

## 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
• Reviewing of study records and source documentation verification in accordance with the monitoring plan

# 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013 and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject

compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

## 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and Sponsor policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed

that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

# 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Data Protection Act of 1998 and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps

should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential

### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

# 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Investigator's Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

Case Report Forms will be completed in real time according to the study procedures specified in the study protocol. Case Report Forms should be completed and reviewed and signed as applicable by the Investigator within 3 days of visit completion. Data queries must be

addressed with complete responses within 3 days of generation. JJVC reserves the right to withhold remuneration until these activities are addressed.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

# **21. PUBLICATION**

This study will be registered on ClinicalTrials.gov.

### 22. REFERENCES

- 1. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP): http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 2. ISO 14155:2011: Clinical investigation of medical devices for human subjects Good clinical practice.
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. <a href="http://www.wma.net/en/30publications/10policies/b3/index.html">http://www.wma.net/en/30publications/10policies/b3/index.html</a>.
- 4. United States (US) Code of Federal Regulations (CFR). In <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a> (Ed.).
- 5. Wirth RJ, Edwards M, Henderson M, et al., Development of the Contact Lens User Experience: CLUE Scales. *Optom Vis Sci.* 2016;93(8):801-808.
- 6. Buch J. Senofilcon-based contact lens containing photochromic dye MXP7-1911 in a 1.2% concentration throughout the entire lens with IPA (Control lens), and PG (Test lens) hydration. 2016.
- 7. Buch J. Confirmation of an investigational lens pilot line clinical performance. 2016.
- 9. Stroup, WS. Generalized linear mixed models. 2012, Boca Raton: CRC Press.
- 10. SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC: SAS Institute Inc; 2014.
- 11. SAS Institute Inc. 2016. SAS/STAT® 14.2 User's Guide. Cary, NC: SAS Institute Inc.




| Protocol 6283 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

| Protocol 6283 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|



**Protocol 6283** 

Protocol 6283

# APPENDIX B: PATIENT INSTRUCTION GUIDE

Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

All polismus ubould be suspiked with a copy of the PATIBIT NSTRUCTION GUIDE for these knows. Copies are emilible for download at wew.acuces.com. Feisien is acceptable, perform a silt temp essertivation to sessess adsopate fi-teresticate and recoverately. If it is acceptable, disperses the brown instruction the appear to return in one week for measurement lines dispersing and fully reformation in FATEM MAMM.GMB-TI.

TORIC FILTING GUIDELINES

Altrody most special of the IRDO procedure are latefact to dispers of each

Altrody most special of the IRDO procedure are latefact to dispers of each

To altrody most special of the College and Altrody control and the College and Altrody control are latefact and procedure developed to ALTRODY

The coll from the college and the procedure of the college and and the procedure and the college and and the procedure and the procedure and the college and

In classification designation of the size here, yet let the size here where yet let the size here where the proposition of the size here. Yet let the size here where yet let the size here where the proposition of the size here where the proposition of the size here where the proposition of the size here where the size here where the size here where the size here where the size here the size here where the size where the size here the size here were with the size here the si

where the course is also also 20 invasion that the course (course in the first NAB or the course and the set present lists at 10 in the last the course of the course of the course of the course of the course of the course of present lists at large course desirated as a usual to set the course that present lists at large course desirated as a usual to set the course of the course of the course of the course of the course of the course of set conjuded to deal to present the course of the course of the course desirated set conjuded to deal the course of the course of the course of the set conjuded to deal the course of the course of the course of the set conjuded to deal the course of the course of the course of the set conjuded to deal the course of the course of the course of the set conjuded to deal the course of the course of the course of the set of the course of the course of the course of the course of the set of the course of the set of the course of

After the patient's parkermora under the above condition is correlated, from a disease of parkers and a parker of the patient

A Administration of the control for models daing the riskle weathing per root for models from the control for models of the control for the co

Assessment of Peterson Comments and Comments

Obode the contration of the sain mark. If the following must in this file of Chock of the contration of the sain stand provided to the stand provided of the sain stand provided at the sain stand of the sain stand or of an addition, red-sail ord stalks.

O.D. 250 - 125 - 110 -

Medical control was consistent and an accordance of the control contro 0.0. ± 0.00 km; the content of the c

REPLACEMENT SCHEDULE

(Mill). Not in Superat on calculations the many of the monomentals for an experimental of the calculation of the many of the m

infects and to convener the lecture infinity. The Eige Care Pollomiscod should specified the infectorized or defector by the finite formular monorized chieful information and produced by the finite formular monorized chieful solid to predict physiological by defensived by the Eige Care Pollomiscode loss that florous version.

A control of the control of the inchmint on the point? NEO may an electron.

AD 1.100 to 1.200 to 2.000 to 2.00

A discrete to extractive could be an entirective country. Before the country of t

HOW SUPPLIED
Each state have it supplied in a fed waterst plades package containing before
solver authorize with neeting etter cells from. The plants; package is marked with the
splawing.

LENS CARE DIRECTIONS
in lease as discoord, the fin Care The best or should provide the patient
and department and department and separate in a confirmation and the
antimizer of the provident of

I sharing

\*\*ACMOT CARTIP Less corn, power, demank it nursies, and requision

\*\*ACMOT CARTIP Less corn, power, demank conner, power, demank

\*\*CARTIP CARTIP LESS CARTIP LESS CARTIPLES (CARTIP LESS CORN)

\*\*CARTIP CARTIP LESS CARTIP C

In a service, the control of the con



Outstann & Jahrenn Weiter Cam Composite 2015 In Carealle, Afrience & Jahrenn Her, Stefann Her, Stefann Her, In 1284, Afrience & African Came Inc. In 1284, Afrience & African Meetin Came Inc. Release after Came Inc.

ACLALE CARTS\* and HTDBACLEAR\* are trademant of Johnson & Johnson Weinn Cass Companies.

# MONOVISION FITTING GUIDELINES

Microsinio Needs Assessment sets the assessment of the assessment

Metod 2 Chamins with one all control selections with head authors in since Albor and an experiment of the selection with the controlled of the selection of the selection of the selection of the chamins of the selection of the selection of the selection of the controlled of the selection of the selection of the selection of the Chamins of the selection of the selection of the selection of the controlled of the selection of the selection of the selection of the chamins of the selection of the selection of the selection of particular of the selection of the selection of the selection of 2 therefore the selection of the selection of the selection of 2 therefore the selection of the selection of the selection of 2 therefore the selection of the selection of the selection of 2 therefore the selection of the selection of the selection of 2 therefore the selection of the selection of the selection of 3 therefore the selection of the selection of the selection of 3 therefore the selection of the selection of the selection of 3 therefore the selection of the selection of 3 therefore the selection of the selection of 3 therefore the selection of the selection of 3 therefore the selection of 3 therefore the selection of 4 therefore the selection of 4 therefore the selection of 4 therefore the selection of 4 therefore the selection of 4 therefore the selection of 5 therefore the s

1. visually demonding alkadions such as operating prioritish physicisms markets or performing other potentially hashinus achieves, and
2. othersy actually out of potentially hashinus achieves, and
alke othersy become multi-prioritism of the proposition of the property of the produced model and
achieves for other which commons, offer may require the additional
over-contribit to the well-back.

2. What Demonst Member: A striple on whether property to these one of the control of the contro

When ADD control and the second and

introffication freeze read carefully and keep this information for kindmentainer for kindmentainer. An expension of the texture of ferring placels is interrode for the type Care Professional, but should be made available to patient on upon request.

The Eye Care Professional should provide the patients with the appropriate instructional deading provide the patients with the appropriate instruction that portation is the patients' prescribed instruction and particular

ACUVUE OASYS BRAND CONTACT LENSES

ACUVUE OASYS\* Brand Contact Lenses
ACUVUE OASYS\* Brand Contact Lenses for ASTIGMA
ACUVUE DASYS\* Brand Contact Lenses for PRESBY

senofficon A Bort (hydrophilis) Contact Lense Visibility Thibd with LIV Blocker for Dally and Extended Wear

R 04/TOYE U.S. Federal law sesticts this device as leavest the device

# SYMBOLS KEY

The following symbols may appear on the label or carbon.

| VI | Consult Instructions for Use |
|---|---|
| 1 | Manufactured by or in |
| U | Date of Manufacture |
| 04 | Use By Date (superation date) |
| TOT | Batch Code |
| - | Steelle Using Steam or Dry Heat |
| EKA | Diamotor |
| 36 | Base Curve |
| 0 | Diopter (lens power) |
| E CHI | Oyluder |
| ADS | Avis |
| MAX ADD | New ADD |
| rom | "Low" Neer ADO |
| OUN | "Medium" New ADD |
| HOR | "High" Near ADD |
| 100 | Quality System Certification Symbol |
| 1 | UV-Booking |
| 0 | Fee Plaid for Waste Management |
| 40 X | CAUTION: U.S. Federal law restricts this device to<br>sale by or on the order of a loanned practitionsr |
| 9, | Lens Orientation Correct |
| 0 | Lens Crientation Incoract Lans Inside Out |

Discord Date on Multi-Purpose Solution Bottle Instructions for Use

Decard any remaining solution althe the recommended time period included on the bodie of malicyapose solution used for districting and mosking the contact lenses.

The Discord Date refers to the time that the pollect can suitely use cor firm care product after the bottle has been opened. It is not the same explaint date, which is the had date that the product is still effective it is opened.

If Margine Conception of the Content of the Content of the Content of Content

These betwee are littled blue using Phacitise Blue Dye #4 to make the letteres mo side for benefits, A benefitiation by about they monorer is used to block Or indicon.

Lear Permission or chrossinelization are lear from 16% in the U/IG approp of 200 mm to

the least that is a between the least of the control of the contro

The political should be abblend to move illum strycter alone to want their known. They have been prescribed to it if their eyes and to correct free values to the degree necessary. Shortly bewas greatly accesses the chance of eye infections.



8.4 et nr. 28 trees
distribute - 4.000 for 0.300 personnests
- 4.500 to - 4.000 for 0.300 personnests
- 6.500 to - 4.000 for 0.300 becoments
- 4.500 to - 4.000 for 0.500 becomments
- 4.500 to - 4.000 for 0.400 personnests
- 4.500 to - 4.000 f

Lemma S. Frakest Dway and the Tye Medidins flow York. 1901; p.50. Span 2-21. Thomas, M. Hattins, Y.M. Sproaf Publisher and Yound Health, CHC Frank, Thomas Theoretisms, Franks.

The second of the second of th

nembaroe characteristics are less than 1% in the UVB narge of 200 ren to and less than 10% in the UVA range of 316 ran to 380 ran for the entire

specificity indicated on product backey by sure highly best and democal
from your better way excepted the sure authors on the production of the production o

An will not contact here. Move up with not recomment to control to the report of the first point and recommend to the report of the repor

vver, clinical studies have not been does to demonstrate that we tocking contact tenses reduces the risk of developing catamots ray distributes. The Epe Gere Professional should be consulted information.

In package (Copyo) grant counts to an included their spiral connection of machine american investor investor and observated in their are design connection of machine interests in the connection of their package

is not a cleaned destination with an ordering and the contact from which contact for the contact for the contact from the con

# ADVERSE REACTIONS the pasteric should be informed that the following problems may occur then wearing contact beness:

The eye may bran, still quality this.

In the eye may bran, still quality this.

The eye may be a second the eye of the e

If the patient reports any problems, he or also about the instructed to MMIDMIT. LYEROYE THE LERS. If the problem or disconfinit stops, the patient should decard the iers and place a new health lens on the eye.

If after inserting the new form, the problem continues, the patient abould be skeeted to MARIDATELY SDACAE THE LIDES AND CONTINUES OR HERE CASE FROMESSORAL.

Vision chunges,

- Loos of Maint,

- Loo of Warner,

- Or Charl gar Problems,

- Or Charl gar Problems,

- Or Problem Strand Charles FOR C

CONTEAUDICATIONS (REACONS NOT TO USE)

The property cents are were for ESPECIATE CRAFFICE, CONT.

We provided youther beautiful for allowing continuous mid
for Active or absolute femalement or whose of the service cheek of the

The continuous femalement or the continuous content of the

The continuous femalement or the continuous content of the continuous content of the continuous content of the content of

for HEMALOUS CONFIGURATION of the Configuration of

# A LOCKWARE AND EXECUTED RELIEF. A RECEIVED WE WAS CONTRICIONED TO CONTRICION (I.G., 10) British ground, by the was of control and out of control a

GENERAL FITTING GUIDELINES
A Priser Solective
Release selected to may three house should be chosen bened once

- Matheritectus ware ferone

- Margin (so decent regarding feros word core

- General levels

- Allath to consume the most cone for the ferone

- Allath to conformated the risk and benefits of leros were

- Allath to conformated the risk and benefits of leros were

2. Others of a file limital area or more of the behaving then behaving the Affe file of the straint and Affe file of the straint and the strai

2. Otherin of a Steep Effect and A A three firstly for may what he can cross of the following described in authorized moment with the back conjugate to be absolute and model when profession he may depend with the house of the first is pulped into a firstly is back in the degree of the papers.

ratio total construction is purport to be fast or attempting the all and admissible, should be should be not extensively distributed of death farm. The farm and bed at mose freely aftern manipulated of deaths for market has a recorded contracted position to these relationships. In contracted above, particular for farm up, the form in filting sightly as degerented to the patient.

Profession with other most the above calcular absolutes the provision with construction.

By the financial activities of the provision of the construction of the cons

# APPENDIX D: CLINICAL TECHNICAL PROCEDURES (CTP)

| Limbal and Conjunctival (Bulbar) Redness |
|-------------------------------------------------------------|
| Expanded Sodium Fluorescein Corneal Staining |
| Lens Fitting Characteristics |
| Subject Reported Ocular Symptoms/Problems |
| Front and Back Surface Lens Deposit Grading Procedure |
| Determination of Distance Spherocylindrical Refractions |
| Biomicroscopy Scale |
| Distance and Near Visual Acuity Evaluation |
| Distance logMAR Visual Acuity Measurement Procedure |
| Patient Reported Outcomes |
| Visual Acuity Chart Luminance and Room Illumination Testing |
| qCSF Contrast Sensitivity |
### , LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS
















### EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING










#### LENS FITTING CHARACTERISTICS















### SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS





# FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE







CR-6283, v3.0 Amendment 2.0 Page 3 of 5
JJVC CONFIDENTIAL






# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















### , BIOMICROSCOPY SCALE













## DISTANCE AND NEAR VISUAL ACUITY EVALUATION











## DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE





CR-6283, v3.0 Amendment 2.0
JJVC CONFIDENTIAL



## , PATIENT REPORTED OUTCOMES





# VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING











## qCSF CONTRAST SENSITIVITY















#### APPENDIX E: IRIS COLOR



#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6283, Initial Evaluation of Investigational Lenses Manufactured on a New Production Line

Version and Date: v3.0, Amendment 2.0, 09 August 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to GCP and ICH guidelines, the Declaration of Helsinki, ISO 14155, United States (US) Code of Federal Regulations (CFR), and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |